CLINICAL TRIAL: NCT04865523
Title: Effectiveness of Manual Lymphatic Drainage in Patients With Fibromyalgia
Acronym: EMLDIPWF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CamiloJcUFM
Record Dates: First submitted 2021-04-24; First posted 2021-04-29 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Fibromyalgia
Keywords: Manual Lymphatic Drainage; Randomized clinical trial; Pain
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Lymphatic Drainage (Experimental)
  Interventions: Other: Manual Lymphatic Drainage
- No intervention (No Intervention)

INTERVENTIONS:
Other: Manual Lymphatic Drainage — Manual lymphatic drainage is a technique that through gentle passes facilitates the flow of lymph through manual therapy techniques based on Vodder therapy. This technique is being studied to know its effectiveness in pain and for this reason we want to carry out this research.
  Arms: Manual Lymphatic Drainage

SUMMARY:
Manual Lymphatic Drainage is a widely used technique for lymphedema. However, the analgesic effects of this technique could be potentially useful for managing pain in patients with generalized widespread chronic pain, including patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Women with diagnosis of Fibromyalgia.

Exclusion Criteria:

* Women with heart failure.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — More Frequently
Enrollment: 30 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold | Baseline
  Kg/cm2
Pain pressure threshold | Immediately after the intervention
  Kg/cm2
Pain pressure threshold | Up to 15 days
  Kg/cm2

SECONDARY OUTCOMES:
Visual Analogue Scale | Baseline
  0-10
Visual Analogue Scale | Immediately after the intervention
  0-10
Visual Analogue Scale | Up to 15 days
  0-10

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Antonio Valera-Calero, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No